CLINICAL TRIAL: NCT03501693
Title: A Multi-Reader Multi-Case Controlled Clinical Trial to Evaluate the Comparative Accuracy of the Fujifilm DBT Plus S-View Versus FFDM Alone in the Detection of Breast Cancer - A Pivotal Study
Brief Title: Fujifilm DBT Plus S-View Versus FFDM Alone in the Detection of Breast Cancer - A Pivotal Study
Status: Completed | Type: Observational
Sponsor: Fujifilm Medical Systems USA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FMSU2017-002B
Record Dates: First submitted 2018-04-02; First posted 2018-04-18 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- DBT plus S-View: Breast images utilizing DBT plus S-View
  Interventions: Device: DBT plus S-View
- FFDM alone: FFDM alone images
  Interventions: Device: FFDM Alone

INTERVENTIONS:
Device: DBT plus S-View — DBT plus S-View images
  Groups: DBT plus S-View
Device: FFDM Alone — FFDM alone images
  Groups: FFDM alone

SUMMARY:
The purpose of the pivotal reader study is to assess the comparative accuracy of Fujifilm DBT plus S-View versus FFDM in the detection of breast cancer.

DETAILED DESCRIPTION:
This clinical research is a retrospective, pivotal, multi-reader, multi-case (MRMC) study with an enriched sample of 300 breast screening or diagnostic cases which were selected from the library of mammograms collected under Fujifilm protocol FMSU2013-004A (all subjects previously provided written informed consent agreeing their image data and supporting documentation could be used for future research and investigations). Approximately 18 qualified radiologists will independently perform two reads on all (approximately 300) cases. Each reader will read each case both as a FFDM read, and a DBT plus S-View read on the ASPIRE Bellus II workstation.

As its primary endpoint, this study is designed to evaluate whether the area under the receiver operating characteristic (ROC) curve (AUC) based on probability of malignancy (POM) scores and requiring correct lesion localization is statistically non-inferior for DBT plus S-View versus FFDM.

ELIGIBILITY:
Inclusion Criteria:

* •Female subjects participating in FMSU2013-004A protocol with known clinical status

Exclusion Criteria:

* •Female subjects that did not have known clinical status in FMSU2013-004A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This is a reader study utilizing retrospectively collected breast images acquired under Fujifilm protocol FMSU2013-004A.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Uzenoff, Study Director — Fujifilm Medical Systems USA, Inc.
Locations (1):
- International HealthCare, LLC, Norwalk, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a retrospective, multi-reader multi-case reader study. 18 radiologist readers read all 300 cases (half FFDM and half DBT plus S-View reads) at each of 2 visits which were separated by a memory washout period of approximately 4 weeks. Images were previously acquired under Fujifilm protocol FMSU2013-004A.
Groups:
- DBT Plus S-View, Then FFDM Only: Readers will read half of the DBT plus S-View images followed by half of the FFDM only images at each of 2 sessions. There was a four week memory washout period between the 2 sessions.
- FFDM Only, Then DBT Plus S-View: Readers will read half of the FFDM images followed by half of the DBT plus S-Viewonly images at each of 2 sessions. There was a four week memory washout period between the 2 sessions.
Period: First Reading Session
Arm/Group | DBT Plus S-View, Then FFDM Only | FFDM Only, Then DBT Plus S-View
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0
Period: 4 Week Memory Washout Period
Arm/Group | DBT Plus S-View, Then FFDM Only | FFDM Only, Then DBT Plus S-View
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0
Period: Second Reading Session
Arm/Group | DBT Plus S-View, Then FFDM Only | FFDM Only, Then DBT Plus S-View
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DBT Plus S-View and FFDM Alone: 300 retrospectively collected breast images to be reviewed (both DBT plus S-View and FFDM alone for all 300 images)
Arm/Group | DBT Plus S-View and FFDM Alone
Number analyzed (Participants) | 300
Age, Customized [Mean (Standard Deviation); unit: years]
  Particant Age Mean | 56.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 300
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 260
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 270
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 300

OUTCOME MEASURES:

1. Primary Outcome: Compare Per Subject AUC: DBT Plus S-View Versus FFDM
Description: Average of each radiologist reader's ROC (receiving operating characteristic curve) based on per-subject POM (probability of malignancy) scores requiring correct lesion localization. A ROC curve is a plot of Sensitivity versus 1-Specificity and is a summary of diagnostic performance of a device or clinician. The reader will first record whether there are mammographic findings and an initial BI-RADS assessment of 0, 1, or 2. If the answer to this question is "no" the reader will be asked to confirm for this case: a BI-RADS assessment category of 1 or 2, a Probability of Malignancy (POM) score following the POM guidance provided in the protocol, and recall decision of "no". If the reader answers "yes" to whether there are mammographic findings, the reader will be asked to confirm an initial BI-RADS assessment category of 0, and will then provide detailed information on each suspicious finding (up to three findings) and the decision whether or not to recall the subject.
Time Frame: 4 weeks
Population: Retrospective images used from Fujifilm protocol FMSU2013-004A. All readers read the same 300 images in their own randomized order during 2 sessions (they read half of each modality at each session which were separated by a 4 week washout period).
Measure: Mean (Standard Error); unit: Probability
Arm/Group | DBT Plus S-View | FFDM Alone
Number analyzed (Participants) | 300 | 300
Probability | 0.794 (0.032) | 0.764 (0.035)

2. Secondary Outcome: Compare Per-subject Average Recall Rate for All Non-cancer Cases for DBT Plus S-View Versus FFDM
Description: Based on recall rate for all non-cancer cases for DBT plus S-View versus FFDM, using non-inferiority margin delta = 0.05. The reader will first record whether there are mammographic findings and an initial BI-RADS assessment of 0, 1, or 2. If the answer to this question is "no" the reader will be asked to confirm for this case: a BI-RADS assessment category of 1 or 2, a Probability of Malignancy (POM) score following the POM guidance provided in the protocol, and recall decision of "no". If the reader answers "yes" to whether there are mammographic findings, the reader will be asked to confirm an initial BI-RADS assessment category of 0, and will then provide detailed information on each suspicious finding (up to three findings) and the decision whether or not to recall the subject, as well as overall POM score and BI-RADS assessment category.
Time Frame: 4 weeks
Population: 240 non-cancer cases evaluated out of 300 total cases acquired under Fujifilm protocol FMSU2013-004A.
Measure: Mean (Standard Error); unit: Proportion of cases correctly recalled
Arm/Group | DBT Plus S-View | FFDM Alone
Number analyzed (Participants) | 240 | 240
Proportion of cases correctly recalled | 0.342 (0.026) | 0.415 (0.027)

3. Secondary Outcome: Compare Per-subject Average Recall Rate for DBT Plus S-View Versus FFDM for All Cancer Cases
Description: Based on recall rate for all cancer cases for DBT plus S-View versus FFDM, using non-inferiority margin delta = 0.10. The reader will first record whether there are mammographic findings and an initial BI-RADS assessment of 0, 1, or 2. If the answer to this question is "no" the reader will be asked to confirm for this case: a BI-RADS assessment category of 1 or 2, a Probability of Malignancy (POM) score following the POM guidance provided in the protocol, and recall decision of "no". If the reader answers "yes" to whether there are mammographic findings, the reader will be asked to confirm an initial BI-RADS assessment category of 0, and will then provide detailed information on each suspicious finding (up to three findings) and the decision whether or not to recall the subject, as well as overall POM score and BI-RADS assessment category.
Time Frame: 4 weeks
Population: 60 cancer cases were read (out of the total of 300 cases) from the previously acquired Fujifilm FMSU2013-004A acquisition study.
Measure: Mean (Standard Error); unit: Proportion of cases correctly recalled
Arm/Group | DBT Plus S-View | FFDM Alone
Number analyzed (Participants) | 60 | 60
Proportion of cases correctly recalled | 0.679 (0.048) | 0.643 (0.049)

4. Secondary Outcome: Compare Per-subject Average Sensitivity for DBT Plus S-View Versus FFDM
Description: Based on forced BI-RADS scores requiring correct lesion localization, using non-inferiority margin delta = 0.10. The reader will first record whether there are mammographic findings and an initial BI-RADS assessment of 0, 1, or 2. If the answer to this question is "no" the reader will be asked to confirm for this case: a BI-RADS assessment category of 1 or 2, a Probability of Malignancy (POM) score following the POM guidance provided in the protocol, and recall decision of "no". If the reader answers "yes" to whether there are mammographic findings, the reader will be asked to confirm an initial BI-RADS assessment category of 0, and will then provide detailed information on each suspicious finding (up to three findings) and the decision whether or not to recall the subject, as well as overall POM score and BI-RADS assessment category.
Time Frame: Four weeks
Population: Sensitivity was analyzed in 60 cancer cases.
Measure: Mean (Standard Error); unit: Probability
Arm/Group | DBT Plus S-View | FFDM Alone
Number analyzed (Participants) | 60 | 60
Probability | 0.679 (0.048) | 0.643 (0.049)

ADVERSE EVENTS:
Time Frame: approximately 5 weeks
Description: There were no AE's expected for this study, as it was a radiologist reader study utilizing retrospective imaging. No study subjects were on-site for this retrospective review. No Adverse Events to report.
Arm/Group | DBT Plus S-View | FFDM Alone
All-Cause Mortality (participants affected / at risk) | 0/300 | 0/300
Serious Adverse Events (participants affected / at risk) | 0/300 | 0/300
Other Adverse Events (participants affected / at risk) | 0/300 | 0/300

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT03501693/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT03501693/SAP_001.pdf